CLINICAL TRIAL: NCT01261871
Title: Intraocular Pressure During Robotic Prostatectomy, Laparoscopic Surgery, and Open Exploratory Laparotomy
Brief Title: Intraocular Pressure During Robotic Assisted Laparoscopic Procedures Utilizing Steep Trendelenburg Positioning
Status: Completed | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NMCSD.2008.0045
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Robotic laparoscopic prostatectomy: Patients who are undergoing primary surgical treatment for a diagnosis of prostate operatively will be enrolled. IOP will be measured throughout the case to assess for change. The various techniques employed for a radical prostatectomy will be compared. Patients undergoing RRP (open surgery) will act as controls. Those undergoing LRP (minimally invasive surgery) will be compared with the control group to assess for differences in IOP that may result from the different approaches. three arms will be used for the comparison: open, laparoscopic intraperitoneal approach), and laparoscopic (extraperitoneal approach).

SUMMARY:
The purpose of this study is to measure pressures within the eye (during surgery to remove the prostate or abdominopelvic masses) as the body position required for these laparoscopic procedures has been associated with increases in pressure within the eye.

DETAILED DESCRIPTION:
The National Cancer Institute estimates that 218,890 new cases of prostate cancer will have been diagnosed in 2007. The three most commonly chosen options for localized prostate cancer are radical prostatectomy (RP), external radiation therapy (XRT), and interstitial brachytherapy (BT). A variety of surgical approaches are available, including open, laparoscopic, and robotic prostatectomy. With the current trend towards "minimally invasive" techniques, laparoscopic prostatectomy (LP) and, in particular, robotic assisted LP are on the rise. Since gaining FDA approval in 2001, the robotic procedure has gained over 1/3 of the market share. Preliminary data suggests this number may now have grown to over 50% of all prostatectomies for cancer performed in the United States.

The minimally invasive procedures offer some advantages relative to the open alternative: smaller incisions, improved pain control, decreased blood loss, and faster recovery have been well documented. Cancer specific and quality of life (sexual function, continence) outcomes will need more long term evaluation before definitive advantages with the minimally invasive techniques are stated. Furthermore, there are potential risks with these minimally invasive methods that have not been fully elucidated.

During a laparoscopic or robotic prostatectomy, patients are subjected to a marked Trendelenberg position throughout the majority of the procedure. The effect of body positioning has been shown previously to affect intraocular pressure (IOP). However, the effect of surgical positioning on IOP during prostatectomies has not been well studied and is not definitively known. Anecdotal reports of postoperative vision loss following robotic assisted laparoscopic prostatectomy have surfaced thus further research is required to study the effect that these procedures for prostate cancer may have on IOP and vision.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients choosing to undergo surgical treatment for prostate cancer

Exclusion Criteria:

* Prior treatment of prostate cancer by any means
* History of glaucoma, macular degeneration, or diabetic retinopathy
* History of eye trauma/injury
* History of non-refractive eye surgery
* Allergy to topical anesthetic (this will be used during the eye exam)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing primary radical prostatectomy for the diagnosis of prostate cancer at Naval Medical Center San Diego.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Effect of radical prostatectomy technique on intraocular pressure. | 30 days post surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Brian K Auge, M.D., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- United States Naval Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No